CLINICAL TRIAL: NCT02018328
Title: The Impact of Addition of Curcumin for 10 Days Triple Therapy, on the Eradication Rate of Helicobacter Pylori Infection
Acronym: CurHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gingold Belfer Rachel (Other)
Responsible Party: Sponsor-Investigator, Gingold Belfer Rachel, MD, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc137511
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Positivity for Helicobacter Pylori
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple therapy, helicobacter pylori (No Intervention)
- triple therapy+curcumin helicobacter pylori (Experimental): Curcumin will be added to the regular triple therapy
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin
  Arms: triple therapy+curcumin helicobacter pylori

SUMMARY:
Background and Aims

* H.pylori is a common human pathogen by which almost 50% of the world population is infected. According to the accepted guidelines, once H.pylori infection has been diagnosed,first line therapy with three drugs should be given. The triple treatment includes proton-pump-inhibitor-clarithromycin-amoxicillin but its eradication rate is only 70-80%.
* Curcumin has many beneficial merits and it was also been demonstrated to be efficient in inhibition of H.pylori infection, in vitro.Therefore we aim to investigate whether addition of Curcumin to the standard triple therapy will increase the eradication rate of H.pylori infection.

Methods

* 150 consecutive patients that will undergo esophagogastroscopy in our Gastroenterology department and will be positive for H.pylori according to urease test and then by gastric biopsy, will be included. The patients will be randomized to two different treatments, according to binomial distribution. 75 patients will be treated with the standard triple therapy for 10 days and the other 75, will be treated for 10 days, with triple therapy combined with Curcumin that will be given three times a day.
* During the treatment the patients will complete an adverse effect's questionnaires. 6 weeks after the completion of the treatment the patients will undergo urea breath test to confirm eradication. Patients will be asked to avoid antibiotics, bismuth compounds or proton-pump-inhibitor until the second urea-breath-test.
* We will compare the eradication rate and the adverse effects between the two groups by using SPSS

ELIGIBILITY:
Inclusion Criteria:

* positivity for Helicobacter pylori by urease test and gastric biopsy

Exclusion Criteria:

* prior treatment for H. pylori
* allergy to penicillin
* gastric outlet obstruction
* pregnancy or breast feeding
* inability to understand the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Urea breath test | 6 weeks after the completion of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Foryst-Ludwig A, Neumann M, Schneider-Brachert W, Naumann M. Curcumin blocks NF-kappaB and the motogenic response in Helicobacter pylori-infected epithelial cells. Biochem Biophys Res Commun. 2004 Apr 16;316(4):1065-72. doi: 10.1016/j.bbrc.2004.02.158. PMID 15044093